CLINICAL TRIAL: NCT07115602
Title: Retrospective Multi-expert Diagnostic Imaging Evaluation of Pelvic Ring Injuries: Methodology for Transferring Large DICOM Data Volumes to Remote Experts, and Survey Designed to Isolate Information Obtained From Different Imaging Modalities
Brief Title: Methodology to Transfer High Volumes of Data for Distant Expert Radiographic Evaluation of Pelvic Ring Injuries
Status: Completed | Type: Observational
Sponsor: Axel Gamulin (Other)
Responsible Party: Sponsor-Investigator, Axel Gamulin, Dr Axel GAMULIN, MD, PD, CC, FMH, Senior Staff Surgeon, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Other Study IDs: VMOO_MDThesis_M_&_M
Record Dates: First submitted 2025-07-16; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Pelvic Ring Injury
Keywords: classification; assessment; computed tomography; stability; pelvic belt; pelvic ring injury; standard anteroposterior radiograph

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pelvic ring injury patients with operative management within 3 weeks from injury: Pelvic ring injury patients with operative management within 3 weeks from injury

SUMMARY:
The aim of this retrospective cohort study based on a prospectively filled registry was to determine whether standard anteroposterior pelvic radiographs with and without pelvic binder provide valuable information on pelvic ring injury anatomy and stability when compared to computed tomography images alone. The ultimate goal was to improve the management of these injuries in both emergency and definitive treatment.

DETAILED DESCRIPTION:
At the core of the study was a stepwise pelvic imaging evaluation of pelvic ring injury patients by a panel of international pelvic trauma experts. The assessment was conducted in 3 sequential steps:

1. Review of computed tomography images alone.
2. Addition of a standard anteroposterior pelvic radiograph with a pelvic binder.
3. Addition of a standard anteroposterior pelvic radiograph without a pelvic binder.

At each step, experts independently classified the injury (Arbeitsgemeinschaft für Osteosynthsesfragen / Orthopaedic Trauma Association and Young and Burgess classifications), assessed mechanical stability and recommended definitive treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1) admission to the author's institution between January 2012 and December 2023;
* 2) high-energy pelvic ring injury involving a non-pathologic pelvis (i.e., no prior injury, pathology, or surgery compromising image interpretation), surgically treated within three weeks of injury;
* 3) age ≥18 years at the time of trauma.

Exclusion Criteria:

* 1) imaging acquired after any kind of surgical stabilization (i.e. emergent external fixation), which could bias injury assessment;
* 2) incomplete imaging dataset, defined as the absence of any of the following: pelvic computed tomography, standard anteroposterior pelvic radiograph with pelvic binder, and standard anteroposterior pelvic radiograph without pelvic binder;
* 3) poor image quality, including incomplete pelvic coverage, computed tomography slice thickness >2 mm, motion artifacts, or incompatibility with the image viewer used for the study;
* 4) documented (written or verbal) refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult pelvic ring injury patients operatively treated within 3 weeks from injury
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Arbeitsgemeinschaft für Osteosynthesefragen / Orthopaedic Trauma Association (AO/OTA) classification | From enrollment to the end of primary injury evaluation at day 1
  Each expert determines the AO/OTA classification of the pelvic ring injury presented by the patient (total = 28 pelvic ring injuries in 28 patients) following a 3 steps sequential imaging evaluation:
  1. Review of computed tomography images alone;
  2. Addition of a standard anteroposterior pelvic radiograph with a pelvic binder;
  3. Addition of a standard anteroposterior pelvic radiograph without a pelvic binder.
  Each one of the 3 provided classifications is recorded and compared to determine if standard anteroposterior pelvic radiographs (with and without a pelvic binder) add value to the information gained with computed tomography images alone in terms of injury classification.
Young and Burgess classification | From enrollment to the end of primary injury evaluation at day 1
  Each expert determines the Young and Burgess classification of the pelvic ring injury presented by the patient (total = 28 pelvic ring injuries in 28 patients) following a 3 steps sequential imaging evaluation: 1) Review of computed tomography images alone; 2) Addition of a standard anteroposterior pelvic radiograph with a pelvic binder; 3) Addition of a standard anteroposterior pelvic radiograph without a pelvic binder. Each one of the 3 provided classifications is recorded and compared to determine if standard anteroposterior pelvic radiographs (with and without a pelvic binder) add value to the information gained with computed tomography images alone in terms of injury classification.
Pelvic ring mechanical stability assessment | From enrollment to the end of primary injury evaluation at day 1
  Each expert determines the mechanical stability of the pelvic ring injury (pelvic ring fully stable, pelvic ring horizontally unstable, pelvic ring fully unstable) presented by the patient (total = 28 pelvic ring injuries in 28 patients) following a 3 steps sequential imaging evaluation: 1) Review of computed tomography images alone; 2) Addition of a standard anteroposterior pelvic radiograph with a pelvic binder; 3) Addition of a standard anteroposterior pelvic radiograph without a pelvic binder. Each one of the 3 provided assessments is recorded and compared to determine if standard anteroposterior pelvic radiographs (with and without a pelvic binder) add value to the information gained with computed tomography images alone in terms of mechanical stability assessment.
Surgical fixation plan | From enrollment to the end of primary injury evaluation at day 1
  Each expert determines the surgical fixation plan (no fixation needed, anterior fixation only, posterior fixation only, lumboelvic fixation only, anterior and posterior fixation, anterior and lumbopelvic fixation) for the pelvic ring injury presented by the patient (total = 28 pelvic ring injuries in 28 patients) following a 3 steps sequential imaging evaluation: 1) Review of computed tomography images alone; 2) Addition of a standard anteroposterior pelvic radiograph with a pelvic binder; 3) Addition of a standard anteroposterior pelvic radiograph without a pelvic binder. Each one of the 3 provided plans is recorded and compared to determine if standard anteroposterior pelvic radiographs (with and without a pelvic binder) add value to the information gained with computed tomography images alone in terms of surgical fixation planning.

IPD SHARING:
Plan to Share IPD: Yes
De-identified radiographic images of the pelvis (computed tomography scanners, standard anteroposterior radiographs with and without pelvic binder)
Supporting Information: Study Protocol
Time Frame: 01.01.2025 for 6 months
Access Criteria: A panel of 8 international pelvic trauma experts was assembled based on their demonstrated expertise in the field and active involvement in relevant academic societies. These 8 experts will receive de-identified radiographic images to classifiy the injuries, evaluate pelvic stability and propose a treatment plan. No other patient data will be shared with the experts.